CLINICAL TRIAL: NCT00943410
Title: Phase II Trial of Herceptin Concurrent With External Beam Radiation Following Neoadjuvant Chemotherapy for the Treatment of HER2 Over-Expressing Breast Cancer
Brief Title: Trastuzumab and External Beam Radiation Therapy in Treating Women With Stage III or Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 9925; CDR000649128 (Other: PDQ); NCT00006109 (obsolete NCT alias)
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: HER2-positive breast cancer; inflammatory breast cancer; recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical Candidate (Active Comparator): After 5 consecutive weeks of treatment with Radiation and Herceptin, these subjects will receive mastectomy excision
  Interventions: Radiation: external beam radiation therapy; Drug: Herceptin
- Non-Surgical Candidate (Active Comparator): After 5 weeks of consecutive treatment with radiation and herceptin, these subjects will not be eligible for surgery. They will continue with radiation and herceptin for an additional 2 weeks.
  Interventions: Radiation: external beam radiation therapy; Drug: Herceptin

INTERVENTIONS:
Radiation: external beam radiation therapy — Radiation therapy will consist of 50Gy in 2Gy fractions to the breast/chest wall and regional lymphatics for 5 consecutive days up to 5 weeks for surgical candidates and 7 weeks for non-surgical candidates
Drug: Herceptin — Patients who are already receiving weekly Herceptin® will continue weekly Herceptin®, 2mg/kg IV on day 1 of each week of radiotherapy. Patients who have not been receiving weekly Herceptin® as a component of systemic therapy will begin Herceptin® one week prior to beginning radiotherapy with a loading dose of 4mg/kg followed by weekly Herceptin® at 2mg/kg on day 1 of each week of radiotherapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy uses high-energy x-rays to kill tumor cells. Trastuzumab may make tumor cells more sensitive to radiation therapy. Giving trastuzumab together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving trastuzumab together with external beam radiation therapy works in treating women with stage III or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the tolerability of trastuzumab (Herceptin®) and concurrent external beam radiotherapy in women with HER2-overexpressing stage III or IV breast cancer.

Secondary

* Determine the pathologic response rate in patients treated with this regimen.
* Determine the locoregional recurrence rate (as site of first recurrence or any recurrence) and time to locoregional recurrence in patients treated with this regimen.
* Determine the time to local progression in patients (who are deemed to be non-surgical candidates) treated with this regimen .

OUTLINE: This is a multicenter study.

Patients receive trastuzumab IV over 30-90 minutes once a week for 5 weeks. Patients also undergo external beam radiotherapy once daily 5 days a week for 5 weeks.

Three weeks after the completion of trastuzumab and radiotherapy, patients undergo surgical evaluation. Patients deemed to be surgical candidates undergo surgery. Patients deemed to be non-surgical candidates continue to receive trastuzumab and external beam radiotherapy for 2 additional weeks.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* invasive primary carcinoma of the breast by fine-needle aspiration, core needle biopsy, or incisional biopsy
* Excisional biopsy is not allowed
* Stage III or IV disease (clinical and radiographic staging), including any of the following:

  * Any T with N2 disease (metastasis to ipsilateral axillary lymph nodes fixed to one another or other structures) or N3 disease (metastasis to ipsilateral internal mammary lymph nodes)
  * T4, any N disease
  * Inflammatory disease
  * Supraclavicular and/or infraclavicular adenopathy
  * Distant metastasis with measurable disease in the breast or lymph nodes
* HER2-overexpressing tumor
* Measurable or evaluable disease
* Residual locoregional disease after completion of neoadjuvant chemotherapy OR locoregional recurrent disease
* Synchronous bilateral primary cancers allowed provided the more serious of the two cancers meets staging criteria
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* WBC > 2,000/mm^3
* Platelet count > 50,000/mm^3
* Hemoglobin > 11 g/dL
* Negative pregnancy test
* Fertile patients must use effective contraception
* Radionucleotide ventriculography/LVEF normal OR ≤ 10% asymptomatic decline from baseline after completion of neoadjuvant chemotherapy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy to the breast or regional lymph nodes
* Concurrent participation in neoadjuvant chemotherapy clinical trials allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2000-03; Primary Completion 2006-01 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events | 7 weeks
  Toxicity (adverse events) will be measured and graded using the CTCAE criteria. RTOG acute toxicity criteria will be used to score acute radiation-related toxicity

SECONDARY OUTCOMES:
Pathologic response rate | 5 weeks
  Pathological response will be measured for those subjects who are deemed surgical candidates. Pathologic response will be defined as invasive tumor present pathologically, or complete invasive tumor clearance (pCR), which includes those tumors with no tumor present as well as those tumors with only in situ carcinoma present after all therapy
Locoregional recurrence rate | up to 5 years
  Radiographic response and recurrence rate will captured using RECIST criteria. Subjects will be followed up for 5 years to document recurrence.
Time to locoregional recurrence | Up to 5 years
  Radiographic response and recurrence rate will captured using RECIST criteria. Subjects will be followed up to 5 years to document recurrence
Time to local progression (in patients who are deemed to be non-surgical candidates) | Up to 5 years
  Radiographic response and recurrence rate will captured using RECIST criteria. Disease progression is defined as an increase in the product of two perpendicular diameters of any measured lesion by > 25% over the size at study entry or the appearance of new areas of malignant disease

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Sartor, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center